CLINICAL TRIAL: NCT06312982
Title: A Series of Neoadjuvant Chemoradiotherapy Combined With Immunotherapy for Locally Advanced Rectal Cancer: From a Multicenter Phase II Cohort to a Phase III Randomized Controlled Study
Brief Title: A Series of Neoadjuvant Chemoradiotherapy Combined With Immunotherapy for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University Cancer Hospital & Institute (Other); China-Japan Friendship Hospital (Other); Peking Union Medical College Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Fudan University (Other); Changhai Hospital (Other); RenJi Hospital (Other); Sir Run Run Shaw Hospital (Other); Shandong Provincial Hospital (Other Government); Zhongnan Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sichuan Academy of Medical Sciences (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Hospital of Jilin University (Other); First Hospital of China Medical University (Other); Xijing Hospital of Airforce Medical University (Unknown); Tangdu Hospital-Air Force Medical University (Unknown); The Affiliated Hospital of Qingdao University (Other); Daping Hospital, the Third Military Medical University (Unknown); Tianjin Union Medical Center (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); The Affiliated Tumour Hospital of China Academy of Medical Science (Unknown); Rocket Force Characteristic Medical Center (Unknown); Tianjin Medical University General Hospital (Other); The Second Affiliated Hospital of Naval Medical University (Unknown); West China Hospital (Other); Southern Medical University - Southern Hospital (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Hebei Medical University Fourth Hospital (Other); Sun Yat-sen University (Other); Zhejiang Tumor Hospital (Other); Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (Unknown); Beijing Hospital of the Ministry of Health (Unknown); Queen Mary Hospital, Hong Kong (Other); The University of Hong Kong-Shenzhen Hospital (Other); Taiwan Hexin Cancer Center Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, The professor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFH-niCRT-04
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Rectal Carcinoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The enrolled patients will receive a long course of NCRT (50 Gy / 25f, capecitabine 850-1000 mg / m2, BID, PO, D1-D5, QW) within the first 5 weeks. In regard to tumor immunotherapy, enrolled patients will receive tislelizumab (200 mg, iv) on the first day at week 2,5, and 8 after initiation of radiotherapy. Thereafter, patients will be treated with two 14-day cycles of the CAPOX（Q 3 w; D1 oxaliplatin, 130mg/m2,iv.gtt; D1-D14, capecitabine, 850-1000mg / m2, BID, PO）regimen. Two CAOPX regimens were treated one week apart. Eight to 8-10 weeks after the completion of radiation therapy, patients will undergo multiple examinations, including colonoscopy and MRI. Subsequent treatment options will be determined by each center physician based on their clinical experience.
  Interventions: Drug: Tislelizumab
- Control group (No Intervention): This group required only 5 weeks of NCRT and two 14-day cycles of the CAPOX （Q 3 w; D1 oxaliplatin, 130mg/m2,iv.gtt; D1-D14, capecitabine, 850-1000mg / m2, BID, PO）regimen.

INTERVENTIONS:
Drug: Tislelizumab — Enrolled patients will receive tislelizumab 3 times after initiation of radiotherapy.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of neoadjuvant chemoradiotherapy combined with tirelizumab compared with neoadjuvant chemoradiotherapy alone for neoadjuvant therapy in patients with locally advanced rectal cancer.

The main questions it aims to answer are:

To evaluate the efficacy and safety of neoadjuvant chemoradiotherapy combined with tirelizumab compared with neoadjuvant chemoradiotherapy alone for neoadjuvant therapy in patients with locally advanced rectal cancer To assess rectal or anal retention as well as quality of life. Participants will receive a long course of NCRT (50 Gy / 25f, capecitabine 850-1000 mg / m2, BID, PO, D1-D5, QW) within the first 5 weeks. In regard to tumor immunotherapy, enrolled patients will receive tislelizumab (200 mg, iv) on the first day at week 2,5, and 8 after initiation of radiotherapy. Thereafter, patients will be treated with two 14-day cycles of the CAPOX（Q 3 w; D1 oxaliplatin, 130mg/m2,iv.gtt; D1-D14, capecitabine, 850-1000mg / m2, BID, PO）regimen. Two CAOPX regimens were treated one week apart.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form and volunteered to join the study;
2. .Age: 18-75 years old, male or female;
3. Pathohistologically confirmed rectal adenocarcinoma, along with immunohistochemical results of pMMR or genetic test results of MSS;
4. The baseline clinical stage assessed by MRI was T1-2N1-2M0 or T3N0-2M0, MRF (-), lateral lymph nodes (-);
5. The lower tumor margin is 10cm away from the anal margin;
6. Surgical resection;
7. Ability to swallow tablets normally;
8. ECOG PS 0-1；
9. Have not received any anti-tumor treatment for rectal cancer, including radiotherapy, chemotherapy, surgery, etc.;
10. Plan to undergo surgery after the completion of the neoadjuvant therapy;
11. No contraindications to surgery;
12. Main organ function is normal.

Exclusion Criteria:

1. Previous history of allergy to monoclonal antibodies, any component of tislelizumab,and capecitabine;
2. Previously has received or is receiving any of the following treatments:

   A)Any tumor-specific surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc; B)Treatment with immunosuppressive drugs or systemic hormones within 2 weeks of first use (dose> 10mg / day prednisone or equivalent dose); inhaled or topical steroids and dose> 10mg / day prednisone or equivalent dose of adrenocorticoid replacement in the absence of active autoimmune disease; C)Having received a live attenuated vaccine within 4 weeks before the first use of the study drug; D)Major surgery or severe trauma within 4 weeks before the first use of study drug;
3. History of any active autoimmune or autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (considered after hormone replacement therapy); patients with psoriasis or asthma / allergy in childhood and adults without any intervention, but patients requiring medical intervention with bronchodilators should not be included;
4. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation or allogeneic bone marrow transplantation;
5. Not well controlled cardiac clinical symptoms or disease, including but not limited to: such as (1) grade NYHA II above heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinical meaningful supraventricular or ventricular arrhythmia without clinical intervention or clinical intervention still poor control;
6. Severe infection (Grade CTCAE> 2) within 4 weeks prior to the first use of study drug, Such as severe pneumonia, bacteremia, infection complications requiring hospitalization; Baseline chest imaging indicated the presence of active lung inflammation, presence of symptoms and signs and signs of infection within 14 days prior to the first administration of study drug or need for oral or intravenous antibiotics, Except for the preventive use of antibiotics; Found active tuberculosis infection by history or CT, Or those with a history of active tuberculosis infection within 1 year prior to enrollment, Or those with a history of active tuberculosis infection more than 1 year ago but without formal treatment;
7. Presence of active hepatitis B (HBV DNA 2000 IU / mL or 104copies / mL), hepatitis C (positive for hepatitis C antibody, and HCV RNA above the lower limit of detection of the analytical method);
8. A diagnosis of other malignancies within 5 years prior to the first use of study drug, unless a malignancy with low risk of metastasis or death (5-year survival> 90%), such as adequately treated skin basal cell carcinoma or squamous cell carcinoma in situ, are considered;
9. Women in pregnancy or lactation;
10. Other factors, as judged by the investigator, may lead to forced termination of the study, such as other serious illness (including mental illness), alcohol, substance abuse, family or social factors, which may affect the safety or compliance of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
CR | pCR :within 10 days after surgery;cCR :13 weeks after radiotherapy begins
  complete response rate=(number of pathological complete responses + number of clinical complete responses)/total number of patients

SECONDARY OUTCOMES:
AE rate | during treatment
  Adverse event rate
NAR score | within 10 days after surgery
  Neoadjuvant rectal（NAR）score：It is based on the scoring criteria of preoperative treatment
ORR | within 10 days after surgery
  objective response rate
  objective response rate
  objective response rate
  objective response rate
OPR | immediately after surgery
  organ preservation rate
  organ preservation rate
  organ preservation rate
immune-related adverse event rate | up to 3 weeks after using tislelizumab
  adverse event rate that is deemed to be associated with tislelizumab

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality